CLINICAL TRIAL: NCT06517329
Title: From Scrubs to Scars: Understanding Bullying Experiences Among Alexandria Faculty of Medicine Students
Brief Title: Bullying Experiences Among Alexandria Faculty of Medicine Students
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: 0305379, IRB NO: 00012098 FWA
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Bullying
Keywords: Bullying, Medical students, learning environment
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study was conducted at Faculty of Medicine, Alexandria to study the prevalence, types and consequences of bullying among medical students. An online survey was distributed among medical students. The data collection continued for two academic years: 2021-2022 and 2022-2023.

DETAILED DESCRIPTION:
A survey based Study was implemented. Questionnaire was used to collect sociodemographic data, exposure to different types if bullying, response and consequences of bullying

ELIGIBILITY:
Inclusion Criteria:

* medical students enrolled at undergraduate or graduate programs of Faculty of medicine who were exposed to bullying

Exclusion Criteria:

* medical students who were not exposed to hullying

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A non-probability sample from all medical students enrolled in undergraduate or graduate programs of Faculty of medicine, Alexandria University, Egypt
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Prevalence | 2021-2023
  Percentage of Students exposed to bullying

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa S. Elhoshy, Principal Investigator — University of Alexandria
Locations (1):
- Faculty of Medicine Alexandria University, Alexandria, Egypt